CLINICAL TRIAL: NCT04768855
Title: A Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of LY3540378 in Healthy Participants
Brief Title: A Study of LY3540378 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: 17793; J3E-MC-EZDA (Other: Eli Lilly and Company)
Record Dates: First submitted 2021-02-23; First posted 2021-02-24 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06-09

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- LY3540378 (Part A) (Experimental): Single ascending doses of LY3540378 administered either intravenously (IV) or subcutaneously (SC).
  Interventions: Drug: LY3540378
- LY3540378 (Part B) (Experimental): Multiple ascending doses of LY3540378 administered SC.
  Interventions: Drug: LY3540378
- LY3540378 (Part C) (Experimental): Multiple ascending doses of LY3540378 administered SC in Japanese Participants.
  Interventions: Drug: LY3540378
- LY3540378 (Part D) (Experimental): Multiple ascending doses of LY3540378 administered SC in Chinese Participants.
  Interventions: Drug: LY3540378
- Placebo (Part A, B, C & D) (Placebo Comparator): Placebo administered either IV or SC.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3540378 — Administered IV or SC.
  Arms: LY3540378 (Part A)
Drug: Placebo — Administered IV or SC.
  Arms: Placebo (Part A, B, C & D)
Drug: LY3540378 — Administered SC.
  Arms: LY3540378 (Part B); LY3540378 (Part C); LY3540378 (Part D)

SUMMARY:
The main purpose of this study is to evaluate the safety and tolerability of the study drug known as LY3540378 in healthy participants following single and multiple doses (Parts A and B) and multiple doses in Japanese (Part C) and Chinese (Part D) healthy participants. Blood tests will be performed to check how much LY3540378 gets into the bloodstream and how long it takes the body to eliminate it. This is a 4-part study and may last up to 70, 113, 113 and 113 days for each participant in Parts A, B, C, and D respectively.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy males or females, as determined by medical history and physical examination.
* Body mass index (BMI) within the range of 19 to 30 kilograms per meter squared (kg/m²)
* For Part C, participants should be first generation Japanese origin.
* For Part D, participants should be first generation Chinese origin.
* Male participants must agree to adhere to contraception restrictions and female participants not of childbearing potential and may include who are infertile due to surgical sterilization (hysterectomy, bilateral oophorectomy, or tubal ligation), or congenital anomaly such as müllerian agenesis or postmenopausal

Exclusion Criteria:

* Participants with troponin I results above the upper reference limit judged to be clinically significant by the investigator
* Diagnosed with orthostatic hypotension defined as a decrease in systolic blood pressure of 20 mm Hg or a decrease in diastolic blood pressure of 10 mm Hg within 3 minutes of standing when compared with blood pressure from the sitting or supine position.
* Have a significant history of or current cardiovascular (for example, myocardial infarction, congestive HF, cerebrovascular accident, venous thromboembolism, etc.), respiratory, renal, gastrointestinal, endocrine, haematological (including history of thrombocytopenia), or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs
* Have obvious clinical signs or symptoms of liver disease, acute or chronic hepatitis biliary and pancreatic disorder
* Have evidence of significant active neuropsychiatric disease as determined by the investigator
* Have received chronic (lasting >14 consecutive days) systemic glucocorticoid therapy in the past year, or have received any glucocorticoid therapy within 1 month before screening
* Have an abnormality in the 12-lead ECG
* Have serum aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >2 × the upper limit of normal (ULN) or total bilirubin (TBL) >1.5 × ULN
* Have a history of acute or chronic pancreatitis or elevation in serum lipase and/or amylase greater than 1.5 × ULN
* Have known allergies to LY3540378 or related compounds
* Have donated blood of >450 mL, or have participated in a clinical study that required similar blood volume drawn within the past 30 calendar days
* Have an average weekly alcohol intake that exceeds 7 units per week, or are unwilling to stop alcohol consumption as required during the study (1 unit = 12 oz or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits)
* Smoke >10 cigarettes per day or the equivalent, or are unable or unwilling to refrain from nicotine
* Allergy to iodine (shellfish allergy)
* Have a history of sensitivity to lithium carbonate

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline up to Day 113
  A summary of SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY3540378 | Predose on Day 1 through Day 113
  PK: Cmax of LY3540378
PK: Area Under the Concentration Versus Time Curve (AUC) of LY3540378 | Predose on Day 1 through Day 113
  PK: AUC of LY3540378

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- Anaheim Clinical Trials, LLC, Anaheim, California, United States
- Lilly Centre for Clinical Pharmacology, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tham LS, Heerspink HJL, Wang X, Verdino P, Saifan CG, Benson EA, Goldsmith P, Wang Z, Testani JM, Haupt A, Sam F, Cherney DZI. Volenrelaxin (LY3540378) increases renal plasma flow: a randomized Phase 1 trial. Nephrol Dial Transplant. 2024 Dec 20;40(1):109-122. doi: 10.1093/ndt/gfae112. PMID 38782726